CLINICAL TRIAL: NCT06814587
Title: Hyperpolarized 13C Pyruvate-MRI and FDG-PET in a Single Exam for the Prognosis of Ischemic Cardiomyopathy
Acronym: FDG PET-HP MRI
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Gaurav Sharma, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2024-0809
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Graft (CABG)
Keywords: Coronary Artery Disease; Hyperpolarized 13C Pyruvate-MRI; FDG-PET; PET-MRI; Myocardial Viability
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Control Group (H): 1.1. Group Description This cohort consists of healthy individuals (n=6) with normal left ventricular ejection fraction (LVEF >50%), no history of coronary artery disease, and no metabolic disorders. Participants will undergo a single session of hyperpolarized 13C pyruvate MRI (HP-13C MRI) and 18F-fluorodeoxyglucose positron emission tomography (FDG-PET) to establish baseline myocardial metabolic and viability parameters.
  Interventions: Diagnostic Test: Hyperpolarized 13C Pyruvate Magnetic Resonance Imaging (HP-13C MRI); Diagnostic Test: [¹⁸F]Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
- Pre-CABG Ischemic Cardiomyopathy (Pre-CABG ICM): 2.1. Group Description This cohort includes patients with ischemic cardiomyopathy (n=6) scheduled for coronary artery bypass grafting (CABG) with LVEF <35%. Participants will undergo preoperative HP-13C MRI and FDG-PET to assess myocardial metabolism and viability prior to revascularization.
  Interventions: Diagnostic Test: Hyperpolarized 13C Pyruvate Magnetic Resonance Imaging (HP-13C MRI); Diagnostic Test: [¹⁸F]Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)
- Post-CABG Follow-up (Post-CABG ICM): 3.1. Group Description This cohort consists of patients post-CABG (n=12), imaged at two follow-up time points: 4-6 months (n=6) and 10-12 months (n=6) after surgery. Participants will undergo repeat HP-13C MRI and FDG-PET to evaluate longitudinal metabolic changes and myocardial functional recovery following revascularization.
  Interventions: Diagnostic Test: Hyperpolarized 13C Pyruvate Magnetic Resonance Imaging (HP-13C MRI); Diagnostic Test: [¹⁸F]Fluorodeoxyglucose Positron Emission Tomography (FDG-PET)

INTERVENTIONS:
Diagnostic Test: Hyperpolarized 13C Pyruvate Magnetic Resonance Imaging (HP-13C MRI) — HP-13C MRI is a metabolic imaging technique that enables real-time assessment of myocardial substrate utilization by tracking the conversion of hyperpolarized [1-13C] pyruvate to metabolic intermediates such as bicarbonate and lactate. This imaging modality provides insights into oxidative metabolism and mitochondrial function, facilitating the identification of metabolically active and ischemic myocardial regions in patients with ischemic cardiomyopathy.
  Other Names: HP 13C-MRI, Hyperpolarized Carbon-13 Pyruvate MRI
Diagnostic Test: [¹⁸F]Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) — FDG-PET is a molecular imaging technique used to assess myocardial viability by quantifying glucose uptake in cardiac tissue. This method differentiates viable myocardium, which retains metabolic activity, from non-viable scar tissue. FDG-PET is widely used in ischemic cardiomyopathy for viability assessment to guide revascularization decisions.
  Other Names: FDG PET, 18F-FDG PET, Fluorodeoxyglucose PET

SUMMARY:
The goal of this clinical trial is to evaluate a novel imaging approach that combines hyperpolarized 13C pyruvate magnetic resonance imaging (HP-13C-MRI) and [¹⁸F]Fluorodeoxyglucose positron emission tomography (FDG-PET) in a single exam to improve the prognostic assessment of ischemic cardiomyopathy. The main questions this study aims to answer are:

Primary Hypothesis: Can the simultaneous acquisition of HP-13C-MRI and FDG-PET data improve the metabolic, viability, and mechanical function assessment in ischemic cardiomyopathy? Primary Outcome Measure: To determine whether the combined HP-13C-MRI/FDG-PET approach provides better prognostic value for ischemic cardiomyopathy compared to current separate imaging modalities.

Secondary Outcome Measures:

Baseline metabolic and viability profiles in healthy individuals. Correlation of metabolic imaging with clinical outcomes in preoperative patients with low left ventricular ejection fraction (LVEF).

Longitudinal changes in myocardial metabolism post-surgery. Study Design: This is a prospective, non-blinded, single-center study utilizing a hybrid PET-MR scanner for simultaneous imaging.

Participants will be divided into three groups:

Healthy subjects (n=6) with normal LVEF for baseline reference. Preoperative patients (n=6) with low LVEF due to ischemic cardiomyopathy undergoing coronary artery bypass grafting (CABG).

Post-CABG patients (n=6 at 4-6 months, n=6 at 10-12 months) to evaluate post-surgical changes.

Procedures:

Undergo HP-13C-MRI and FDG-PET imaging in a single session. Blood samples for metabolic biomarkers (lactate, pyruvate, triglycerides, insulin, glucose).

Standard clinical cardiac imaging (Echocardiography, SPECT Myocardial Perfusion Imaging).

DETAILED DESCRIPTION:
1. Study Rationale and Significance 1.1. Ischemic Cardiomyopathy and the Need for Advanced Imaging Approaches Ischemic cardiomyopathy (ICM) is a progressive disorder characterized by myocardial dysfunction due to reduced coronary perfusion, most commonly caused by underlying coronary artery disease (CAD) or previous myocardial infarction (MI). The prognosis of ICM remains poor, with high rates of morbidity and mortality despite advances in pharmacologic, interventional, and surgical therapies. A major clinical challenge in managing ICM is the accurate and comprehensive assessment of myocardial viability and metabolic function to guide appropriate revascularization strategies. Traditional imaging techniques, including late gadolinium-enhanced cardiac magnetic resonance imaging (LGE-CMR), single-photon emission computed tomography (SPECT), and dobutamine stress echocardiography, provide structural and functional insights but are limited in their ability to dynamically assess metabolic alterations that precede irreversible myocardial damage.

   1.2. Limitations of Current Imaging Modalities in Assessing Viability and Metabolism Existing non-invasive imaging approaches for myocardial viability assessment rely primarily on anatomical markers of fibrosis, contractile reserve, or static glucose metabolism, requiring multiple imaging sessions with different modalities. These approaches pose several limitations, including discordant results between imaging techniques, increased patient burden due to multiple appointments, and delays in treatment decisions. More importantly, the lack of an integrated imaging strategy limits the ability to assess real-time metabolic adaptations that can predict myocardial recovery potential post-revascularization.

   1.3. The Rationale for a Combined HP-13C MRI and FDG-PET Imaging Approach The proposed study seeks to overcome these limitations by employing a novel integrated metabolic imaging method combining hyperpolarized 13C-pyruvate magnetic resonance imaging (HP-13C-MRI) and [¹⁸F]Fluorodeoxyglucose positron emission tomography (FDG-PET) in a single examination. HP-13C-MRI provides real-time metabolic flux information, allowing direct visualization of substrate utilization and oxidative metabolism, while FDG-PET enables quantification of glucose uptake and viability assessment. By simultaneously acquiring metabolic, viability, and mechanical function data, this hybrid approach has the potential to transform the diagnostic paradigm for ischemic cardiomyopathy.
2. Study Objectives and Hypotheses 2.1. Primary Objective The primary objective of this study is to determine whether simultaneous HP-13C-MRI and FDG-PET imaging can improve the assessment of myocardial viability and metabolic function in ischemic cardiomyopathy compared to current standard imaging approaches.

   2.2. Secondary Objectives

   The secondary objectives include:

   2.2.1. Establishing baseline myocardial metabolism, viability, and mechanical function parameters in healthy subjects using combined HP-13C-MRI and FDG-PET to serve as a reference for subsequent patient cohorts.

   2.2.2. Evaluating metabolic abnormalities in preoperative patients with ischemic cardiomyopathy and low left ventricular ejection fraction (LVEF) to correlate metabolic activity with clinical disease severity and revascularization outcomes.

   2.2.3. Conducting a longitudinal assessment of myocardial metabolism and function following surgical revascularization to determine the predictive value of baseline metabolic imaging for post-surgical myocardial recovery.

   2.3. Primary Hypothesis It is hypothesized that the simultaneous acquisition of metabolic and viability data via HP-13C-MRI and FDG-PET in a single imaging session will provide superior diagnostic accuracy and prognostic value for ischemic cardiomyopathy compared to standard imaging techniques performed separately.

   2.4. Secondary Hypotheses 2.4.1. In healthy individuals with normal myocardial function, HP-13C-MRI and FDG-PET will establish normal metabolic flux patterns, which will differ significantly from those observed in patients with ischemic cardiomyopathy.

   2.4.2. In preoperative patients with ischemic cardiomyopathy, metabolic derangements detected via HP-13C-MRI will correlate with regional glucose uptake on FDG-PET and provide insights into myocardial segments with reversible dysfunction.

   2.4.3. Post-CABG follow-up imaging will demonstrate metabolic improvement in viable myocardial segments, confirming the potential of preoperative metabolic imaging as a predictive tool for post-revascularization myocardial recovery.
3. Study Design and Methodology 3.1. Study Type and Design This is a prospective, single-center, non-blinded translational research study employing a hybrid PET-MR scanner for simultaneous imaging.

   3.2. Study Population and Group Allocation

   A total of 12 human subjects will be enrolled, stratified into three groups:

   3.2.1. Healthy control group (n=6) consisting of individuals with normal LVEF (>50%) to establish baseline metabolic and viability reference values.

   3.2.2. Pre-CABG ischemic cardiomyopathy group (n=6) consisting of patients with reduced LVEF (<35%) undergoing planned coronary artery bypass grafting (CABG).

   3.2.3. Post-CABG follow-up group (n=6 at 4-6 months, n=6 at 10-12 months) consisting of the same pre-CABG cohort undergoing post-surgical follow-up imaging to assess metabolic recovery.

   3.3. Study Procedures 3.3.1. All participants will undergo one or two imaging sessions involving HP-13C-MRI and FDG-PET in a single session using a hybrid PET-MR scanner.

   3.3.2. Participants will undergo blood sampling before and after imaging to measure key metabolic biomarkers, including lactate, pyruvate, triglycerides, insulin, and glucose.

   3.3.3. Clinical cardiac imaging data, including echocardiography, SPECT myocardial perfusion imaging, and invasive coronary angiography, will be collected for correlation with metabolic imaging findings.

   3.4. Imaging Protocol 3.4.1. Hyperpolarized 13C Pyruvate MRI Acquisition 3.4.1.1. Hyperpolarized [1-13C] pyruvate will be dynamically injected, and real-time conversion to metabolic intermediates (bicarbonate and lactate) will be measured.

   3.4.1.2. Cardiac-gated 13C imaging sequences will be used to quantify myocardial metabolic flux, focusing on segmental variations in oxidative metabolism.

   3.4.2. FDG-PET Acquisition 3.4.2.1. FDG uptake will be measured to assess myocardial viability and regional glucose metabolism.

   3.4.2.2. Metabolic activity will be compared across ischemic and non-ischemic myocardial regions.
4. Data Analysis and Statistical Considerations 4.1. Primary Statistical Analysis 4.1.1. HP-13C MRI and FDG-PET data will be analyzed using MATLAB-based reconstruction and analysis pipelines.

   4.1.2. Quantitative metabolic parameters, including bicarbonate-to-lactate ratio and myocardial FDG uptake, will be compared across study groups.

   4.1.3. Statistical significance will be determined using an unpaired t-test (α=0.05, one-tailed) for two-group comparisons and ANOVA/2-way ANOVA for multi-group comparisons.

   4.2. Sample Size Justification 4.2.1. The sample size of 12 subjects (24 imaging sessions) is based on feasibility and prior studies demonstrating significant metabolic differences with HP-13C MRI in small cohorts.

   4.2.2. Power calculations suggest that this sample size will be sufficient to detect clinically relevant differences in myocardial metabolic parameters with an estimated effect size of 1.0 and 80% power at α=0.05.
5. Safety and Risk Considerations 5.1. Radiation Exposure 5.1.1. The combined HP-13C MRI and FDG-PET protocol will result in a radiation exposure of ~10.5 mSv, within acceptable diagnostic limits.

5.1.2. Radiation exposure will be monitored to comply with institutional and regulatory guidelines.

5.2. Adverse Event Monitoring 5.2.1. Subjects will be closely monitored during imaging, with continuous ECG and blood pressure monitoring.

5.2.2. Any adverse events will be reported and managed according to institutional safety protocols.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

* Age between 20-80 years
* Eligible for MRI, PET, and contrast agents (based on institutional screening protocols)
* Scheduled for CABG (for ischemic cardiomyopathy patients)
* Left ventricular ejection fraction (LVEF) ≤ 40% or clinical indication for myocardial viability assessment
* No history of coronary artery disease or diabetes (for healthy controls)
* Negative pregnancy test (for female participants of childbearing potential)

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

* Age <20 or >80 years
* Prior extensive myocardial infarction (defined as >50% transmural scar on viability imaging)
* Contraindications to MRI, PET, or contrast agents (including severe claustrophobia or allergy)
* Pregnant or breastfeeding women
* Severe renal impairment (GFR <30 mL/min/1.73m²)
* Uncontrolled diabetes (HbA1c >9%)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes patients with ischemic cardiomyopathy undergoing CABG and healthy controls to establish metabolic reference values.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Myocardial Metabolic and Viability Assessment via HP-13C MRI and FDG-PET | Baseline imaging at enrollment (pre-CABG, within 30 days before surgery)
  This outcome measures the ability of combined hyperpolarized 13C pyruvate MRI (HP-13C MRI) and FDG-PET in a single imaging session to assess myocardial metabolic function and viability in ischemic cardiomyopathy. Quantitative assessment will include the bicarbonate-to-lactate ratio (HP-13C MRI) and regional FDG uptake (FDG-PET). The prognostic accuracy of these metabolic markers will be compared against standard viability imaging techniques.

SECONDARY OUTCOMES:
Comparison of Myocardial Metabolic Profiles in Healthy vs. Ischemic Cardiomyopathy Patients | Baseline imaging at enrollment (single session within 14 days of consent)
  This outcome evaluates differences in myocardial metabolic parameters (bicarbonate/lactate ratio, FDG uptake) between healthy controls and preoperative ischemic cardiomyopathy patients. The goal is to establish metabolic reference values in healthy myocardium and determine metabolic alterations in ischemic regions.
Longitudinal Changes in Myocardial Metabolism Post-CABG | Follow-up imaging at 4-6 months (±2 weeks) and 10-12 months (±2 weeks) post-CABG.
  This outcome assesses metabolic and functional changes in myocardial segments post-revascularization by evaluating HP-13C MRI and FDG-PET parameters at 4-6 months and 10-12 months post-CABG. Improvement in myocardial oxidative metabolism and glucose uptake will be correlated with functional recovery.
Correlation of Preoperative Metabolic Imaging with Post-Surgical Cardiac Function | LVEF and cardiac function measured at baseline (pre-CABG, within 30 days before surgery), 4-6 months (±2 weeks) post-CABG, and 10-12 months (±2 weeks) post-CABG.
  This outcome investigates whether preoperative metabolic imaging findings predict post-surgical improvement in left ventricular ejection fraction (LVEF) and regional wall motion.

OTHER OUTCOMES:
Feasibility and Reproducibility of Combined HP-13C MRI and FDG-PET in a Single Imaging Session | Assessed at each imaging session (baseline imaging within 14 days of consent, follow-up imaging at 4-6 months and 10-12 months post-CABG).
  This outcome assesses technical feasibility, image quality, and inter-scan reproducibility of HP-13C MRI and FDG-PET acquisition in a single session. Factors evaluated include signal-to-noise ratio (SNR), metabolic quantification precision, and scan duration tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Sharma, PhD, MBA, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No